CLINICAL TRIAL: NCT01555567
Title: Quadriceps Inhibition After ACL Injury: Neuromuscular and Functional Consequences
Brief Title: Electrical Stimulation and Eccentric Exercise for Anterior Cruciate Ligament (ACL) Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Principal Investigator, Riann Palmieri-Smith, Associate Professor, University of Michigan
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ACLNMES; 1K08AR053152-01A2 (NIH)
Record Dates: First submitted 2012-03-06; First posted 2012-03-15 (Estimated); Results first posted 2015-05-14 (Estimated); Last update posted 2015-06-08 (Estimated); Status verified 2015-05

CONDITIONS: Anterior Cruciate Ligament Injury
Keywords: ACL; muscle; quadriceps; strength
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries | interventions — Electric Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Electrical stimulation (Experimental): Subjects placed into this group will undergo electrical stimulation following anterior cruciate ligament reconstruction (ACLr). Subjects will be required to report 2 times per week for 6 weeks following ACLr for electrical stimulation therapy. Electrical stimulation therapy post-reconstruction will commence immediately post-ACLr and end at week 6.
  Interventions: Device: Electrical Stimulation
- Standard of Care (No Intervention): This group will undergo standard ACL rehabilitation
- Eccentric Exercise (Experimental): Subjects placed into this group will undergo eccentric exercise strength training following ACLr. Subjects will be required to report 2 times per week for 6 weeks following ACLr. Eccentric strengthening will begin at week 6 post-ACLr and will end at week 12 post-ACLr.
  Interventions: Other: Eccentric Exercise
- Stimulation and Eccentrics (Experimental): Subjects placed into this group will undergo a combined electrical stimulation and eccentric exercise intervention following ACLr. The electrical stimulation intervention will be delivered immediately following ACLr and will end at 6 weeks post-ACLr. Subjects will receive the electrical stimulation therapy 2 times per week for the first 6 weeks post-ACLr. At six weeks post-ACLr, subjects will begin the eccentric strengthening protocol. Subjects will eccentrically train 2 times per week for 6 weeks. The eccentric strengthening will end at 12 weeks post-ACLr.
  Interventions: Device: Electrical Stimulation; Other: Eccentric Exercise

INTERVENTIONS:
Device: Electrical Stimulation — Electrical stimulation will be delivered 2 times per week
  Arms: Electrical stimulation; Stimulation and Eccentrics
Other: Eccentric Exercise — Eccentric Exercise will be delivered 2 times per week
  Arms: Eccentric Exercise; Stimulation and Eccentrics

SUMMARY:
Quadriceps muscle weakness is a common consequence of ACL injury. This muscle weakness is considered to result from neural inhibition preventing full muscle contraction and is referred to as arthrogenic muscle inhibition (AMI). AMI hinders rehabilitation by preventing gains in strength, increasing the risk of re-injury, and potentially placing patients at risk for chronic degenerative joint conditions. Quadriceps weakness that occurs following ACL injury is also thought to be caused by muscle atrophy which is thought to manifest due to alterations in muscle architecture, selective fiber atrophy or even neural deficits such as AMI. Importantly, interventions that are designed to counter this muscle weakness are required in order to promote long-term knee joint health. Hence, the purpose of the current study is to determine the efficacy of interventions that target quadriceps weakness to improve quadriceps muscle function and biomechanics in patients prior to and following ACL reconstruction. Specifically, the efficacy of neuromuscular electrical stimulation aimed at improving quadriceps neural activity and eccentric exercise intended to minimize quadriceps muscle atrophy will be investigated. The investigators expect that patients who receive the electrical stimulation therapy will demonstrate improvements in quadriceps strength and activation. Furthermore, it is expected that patients who receive both the electrical stimulation and eccentric intervention will demonstrate markedly greater gains in quadriceps strength and activation than patients who receive only the electrical stimulation therapy or standard of care post-surgery. The investigators also hypothesize that the patients who receive the electrical stimulation therapy and/or eccentrics will display knee motion similar to uninjured control subjects.

DETAILED DESCRIPTION:
Neuromuscular electrical stimulation (NMES) has been shown to reduce quadriceps activation failure (QAF) and eccentric exercise has been shown to lessen muscle atrophy post-ACL reconstruction. Given thatthese are two critical components of quadriceps strength, intervention combining these therapies may be effective at reinstituting quadriceps function post-reconstruction. Therefore, the aim of this study is to evaluate the effectiveness of a combined NMES and eccentric exercise intervention to improve the recovery of quadriceps activation and strength post-reconstruction. Patients post ACL-injury will be placed into four treatment groups (NMES and eccentrics; eccentrics only; NMES only, and standard of care) Patients assigned to the NMES and eccentric and the NMES only groups will receive the NMES protocol 2× per week for the first 6 weeks post-reconstruction. MES and eccentric and the eccentrics only groups will receive the eccentric exercise protocol 2× perweek beginning 6 weeks post-reconstruction. Quadriceps activation was assessed via the superimposed burst technique and quantified via the central activation ratio.Quadriceps strength was assessed via maximal voluntary isomeric contractions (Nm/kg). Data will be gathered on three occasions: pre-operative, 12-weeks-post-surgery and at return-to-play.

ELIGIBILITY:
Inclusion Criteria:

* Aged 14-35 years
* Willingness to participate in testing and follow-up as outlined in the protocol
* Scheduled to undergo ACL reconstruction

Exclusion Criteria:

* Previous quadriceps injury
* Inability to provide informed consent
* Pregnant females
* ACL injury sustained more than 48 hours prior to reporting to physician
* ACL injury sustained when not engaged in sports participation (i.e. while engaged in activities of daily living)
* Previous partial ACL tear
* Previous surgery to injured knee
* Total or partial meniscectomy accompanying ACL reconstruction
* Other ligamentous injury accompanying ACL injury

Ages: 14 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 43 (Actual)
Dates: Start 2009-08; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Riann M Palmieri-Smith, PhD, Principal Investigator — University of Michigan
Locations (1):
- MedSport, Ann Arbor, Michigan, United States

REFERENCES:
- [Derived] Lepley LK, Palmieri-Smith RM. Quadriceps Strength, Muscle Activation Failure, and Patient-Reported Function at the Time of Return to Activity in Patients Following Anterior Cruciate Ligament Reconstruction: A Cross-sectional Study. J Orthop Sports Phys Ther. 2015 Dec;45(12):1017-25. doi: 10.2519/jospt.2015.5753. Epub 2015 Oct 15. PMID 26471854

RESULTS

PARTICIPANT FLOW:
Groups:
- Neuromuscular Electrical Stimulation: Subjects placed into this group will undergo neuromuscular electrical stimulation (NMES) following anterior cruciate ligament (ACLr). Subjects will be required to report 2 times per week for 6 weeks following ACLr for NMES therapy. NMES therapy post-reconstruction will commence immediately post-ACLr and end at week 6.
  Neuromuscular Electrical Stimulation: NMES will be delivered 2 times per week
- Combination of NMES and Eccentric Exercise: Subjects placed into this group will undergo a combined NMES and eccentric exercise intervention following ACLr. The NMES intervention will be delivered immediately following ACLr and will end at 6 weeks post-ACLr. Subjects will receive the NMES therapy 2 times per week for the first 6 weeks post-ACLr. At six weeks post-ACLr, subjects will begin the eccentric strengthening protocol. Subjects will eccentrically train 2 times per week for 6 weeks. The eccentric strengthening will end at 12 weeks post-ACLr.
  Neuromuscular Electrical Stimulation: NMES will be delivered 2 times per week
  Eccentric Exercise: Eccentric Exercise will be delivered 2 times per week
Period: 12 Week
Arm/Group | Neuromuscular Electrical Stimulation | Standard of Care | Eccentric Exercise | Combination of NMES and Eccentric Exercise
Started | 12 | 13 | 9 | 9
Completed | 11 | 12 | 8 | 9
Not Completed | 1 | 1 | 1 | 0
Period: Return to Activity
Arm/Group | Neuromuscular Electrical Stimulation | Standard of Care | Eccentric Exercise | Combination of NMES and Eccentric Exercise
Started | 11 | 12 | 8 | 9
Completed | 10 | 10 | 8 | 8
Not Completed | 1 | 2 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Neuromuscular Electrical Stimulation: Subjects placed into this group will undergo NMES following ACLr. Subjects will be required to report 2 times per week for 6 weeks following ACLr for NMES therapy. NMES therapy post-reconstruction will commence immediately post-ACLr and end at week 6.
  Neuromuscular Electrical Stimulation: NMES will be delivered 2 times per week
- Total: Total of all reporting groups
Arm/Group | Neuromuscular Electrical Stimulation | Standard of Care | Eccentric Exercise | Combination of NMES and Eccentric Exercise | Total
Number analyzed (Participants) | 10 | 10 | 8 | 8 | 36
Age, Continuous [Mean (Standard Deviation); unit: years] | 21.8 (4.4) | 18.3 (3.7) | 23.2 (5.4) | 23.2 (6.3) | 21.6 (4.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 5 | 3 | 3 | 13
  Male | 8 | 5 | 5 | 5 | 23
Region of Enrollment [Number; unit: participants]
  United States | 10 | 10 | 8 | 8 | 36
Height [Mean (Standard Deviation); unit: meter] | 1.76 (.1) | 1.73 (.1) | 1.75 (.1) | 1.45 (.6) | 1.67 (.22)
Mass [Mean (Standard Deviation); unit: kg] | 81.65 (22.6) | 75.5 (24.1) | 77.7 (10.4) | 77.8 (16.5) | 78.2 (18.4)
Quadriceps Strength [Mean (Standard Deviation); unit: Nm/kg] | 2.6 (.6) | 2.6 (.6) | 2.8 (1.1) | 2.7 (.8) | 2.67 (.78)
Central Activation Ratio (CAR) [Mean (Standard Deviation); unit: ratio] — CAR = maximal voluntary isometric contraction force / maximal voluntary isometric contractions force + stimulated force
  ratio | 97.4 (3) | 94.9 (5.3) | 95.9 (4.5) | 95.7 (3.5) | 95.9 (4.1)

OUTCOME MEASURES:

1. Primary Outcome: Quadriceps Strength
Time Frame: Time of return to activity (~6 months following surgery)
Measure: Mean (Standard Deviation); unit: Nm/kg
Arm/Group | Neuromuscular Electrical Stimulation | Standard of Care | Eccentric Exercise | Combination of NMES and Eccentric Exercise
Number analyzed (Participants) | 10 | 10 | 8 | 8
Nm/kg | 2.1 (0.6) | 2.1 (0.6) | 2.8 (0.9) | 2.9 (0.6)

2. Secondary Outcome: Central Activation Ratio
Description: CAR = maximal voluntary isometric contractions force / maximal voluntary isometric contractions force + stimulated force
Time Frame: Time of return to activity (~6 months following surgery)
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Neuromuscular Electrical Stimulation | Standard of Care | Eccentric Exercise | Combination of NMES and Eccentric Exercise
Number analyzed (Participants) | 10 | 10 | 8 | 8
ratio | 91.8 (4.6) | 91.8 (9) | 98.1 (1.2) | 97.6 (2.8)

ADVERSE EVENTS:
Arm/Group | Neuromuscular Electrical Stimulation | Standard of Care | Eccentric Exercise | Combination of NMES and Eccentric Exercise
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 0/8 | 0/8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No